CLINICAL TRIAL: NCT00775151
Title: The Objective of This Study Was to Compare the Rate and Extent of Absorption of Ranbaxy Amlodipine 10 mg Tablet to That of Norvasc® 10 mg Tablet After a Single, One Tablet Dose in Fed State Subjects.
Brief Title: Bioequivalence Study of Amlodipine 10mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 50366
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence amlodipine 10 mg tablet under fed conditions
MeSH Terms: interventions — Amlodipine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): amlodipine 10 mg tablet of Ranbaxy
  Interventions: Drug: amlodipine 10 mg tablet
- 2 (Active Comparator): Norvasc® 10 mg tablets
  Interventions: Drug: amlodipine 10 mg tablet

INTERVENTIONS:
Drug: amlodipine 10 mg tablet

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of Ranbaxy amlodipine 10 mg tablet to that of Norvasc® 10 mg tablet after a single, one tablet dose in fed state subjects.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioequivalence study on Amlodipine besylate formulations comparing Amlodipine 10mg tablets of Ranbaxy Laboratories with (Norvasc®, Pfizer Inc USA, in healthy, adult, human, subjects under fed conditions

Enrolled and randomized: 40 each treatment) Drop-outs (withdrew from study): 1 Withdrawals (was dropped from study): 4 Completed: 36

ELIGIBILITY:
Inclusion Criteria:

* Is the individual a healthy, normal adult man and woman who volunteers to participate? ls s/he at least 18 years of age? Is his/her BMI between 19 and 30, inclusive? Is she willing .to avoid pregnancy by abstaining from sexual intercourse with a non-sterile male partner, or by the use one of the following methods: diaphragm + spermicide or condom + spermicide (at least 14 days before dosing), intra- uterine contraceptive device or hormonal contraceptives (at least 4 weeks prior to dosing), or has she been surgically sterile or post-menopausal at least six months prior to entering into the stndy?

  * Is s/he considered .reliable and capable of understanding his/her responsibility and role in the study.
  * Has s/he provided written informed consent?

A no answer to any of the above questions indicated that the individual was ineligible for enrollment

Exclusion Criteria:

* Does the individual have a history of allergy or hypersensitivity to amlodipine? Does s/he have clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his/her safety?
* Does s/he have significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hematopoietic, hepatic, neurological, ongoing infection, pancreatic, or renal diseases that would interfere with the conduct or interpretation of the study or jeopardize his/her safety'?
* Is she nursing?
* Does s/he have serious psychological illness?
* Does s/he have significant h/story (within the past year) or clinical evidence of alcohol or drug abuse? •
* Does s/he have a positive urine drug screen or a positive HIV-1, or hepatitis B or C screen, or a positive pregnancy test? Has s/he consumed grapefruit or grapefruit juice during the 7rday period preceding study initiation?
* Is s/he unable to refrain from the use of alcohol or xanthine-containing foods or beverages during periods beginning 48 hours prior to study drug administration and ending when the last blood sample has been taken in each study period?
* Has s/he used any prescription drug, other than hormonal contraceptives, during the 14-day period prior to study initiation, or any OTC drug during the 72-hour period preceding study initiation?
* Is s/he unable to refrain from the use of all concomitant medications, other than hormonal contraceptives, during the study?
* Has s/he donated or lost blood, or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six week period preceding study initiation?

Has s/he donated plasma during the two week period preceding study initiation? Has s/he received an investigational drug during the 30 day period preceding study initiation? Is s/he a heavy smoker (usually smoking more than 10 cigarettes per day)?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2005-08 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- SFBC Ft. Myers, Inc., Fort Myers, Florida, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm